CLINICAL TRIAL: NCT06797440
Title: The Effect of Dual Tasks of Digital Technology on Cognitive Function and Physical Activity in the Older Adults With Cognitive Frailty - A Randomized Controlled Trial
Brief Title: The Effect of Dual Tasks of Digital Technology on Cognitive Function and Physical Activity in the Older Adults With Cognitive Frailty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Chia Jung Hsieh, Ph.D., RN, Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: C113026
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Frailty
Keywords: Cognitive Frailty; Dual task; Digital technology; Nintendo Switch; Physical activity; Cognition funtion
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of digital technology interventions, it is difficult to blind study caregivers and participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): The experimental group received a dual-task protocol. The intervention activities of the experimental group were cognitive and physical activity training using Nitendo Switch.
  Interventions: Other: Dual tasks of digital technology
- Control group (No Intervention): The control group received usual care.

INTERVENTIONS:
Other: Dual tasks of digital technology — The intervention activities of this study were cognitive and physical activity training using Nintendo Switch twice a week, 60 minutes each time (5 minutes of warm-up and cool-down exercises, 10 minutes of stretching exercises, and 40 minutes of exercise combined with cognitive training) for a total of 8 weeks. train. Both groups filled in basic data (demographics and disease characteristics) and underwent cognitive function measurements and physical activity function measurements at pretest (T0), 4th week (T1), and 8th week (T2).
  Arms: Experimental group

SUMMARY:
Background: Cognitive frailty is a state that combines physical weakness and cognitive impairment. As age increases, the prevalence rate also increases. Older adults with cognitive frailty are prone to falls, limited or degraded physical functions, and are at high risk of becoming disabled. It is an essential predictor of dementia and mortality. There are currently very few randomized controlled trial studies on cognitive frailty abroad. Although there are many related studies on senile frailty in Taiwan, most studies examine cognitive function and physical frailty separately. Since cognitive frailty is reversible, early intervention can delay or prevent the occurrence of cognitive frailty. Therefore, cognitive-motor dual tasks are introduced. For more information, see the effectiveness of dual-tasking in cases of cognitive decline.

Purpose: Goal is to not only explore the feasibility of a motor-cognition dual-task program for elderly individuals with cognitive frailty but also to compare its impact on cognitive and physical function with existing training programs. By doing so, the purpose of this study will be to provide practical insights that can inform the development of effective interventions for this vulnerable population.

Methods: A randomized clinical trial was used to explore the effectiveness of a dual-task intervention program on cognitive function and physical activity in older adults with cognitive frailty. Eligible subjects were recruited through convenience sampling and randomly assigned to two groups. The experimental group used Nintendo Switch to perform dual tasks of motor cognition, while the control group performed regular activities. Twice a week, 60 minutes each time, for eight weeks of training. Both groups completed basic information (demographics, disease characteristics, and lifestyle), cognitive function measurements, and physical activity function measurements in the pre-test (T0) in the 4th week (T1) and 8th week (T2). Cognitive function measurements and physical activity function measurements were performed again. Using SPSS 29.0 as a statistical tool, independent sample t-test and Chi-square test were used to detect the demographic variables, disease treatment variables, living habits, cognitive functions, and physical effects of the two groups-homogeneity of activities. A generalized estimating equation (GEE) was used as a statistical method to process and analyze repeated measurement data. The effects of the inter-group and time interaction on the two groups' cognitive function and physical activity were studied differently.

Expected research results: This study is expected to construct a suitable dual-task program to introduce the role of physical and cognitive function in this group and explore its effectiveness.

DETAILED DESCRIPTION:
Background:

As the population ages, the number of diseases or problems related to old adults is also increasing, among which the problem of frailty is also rising sharply. Scholars define frailty as multiple declines in physiological systems, which lead to the deterioration of body reserve functions, increase the susceptibility to clinical symptoms, and reduce The ability to cope with acute stress, leading to related complications and adverse health outcomes, such as falls, decreased physical activity, cognitive decline, and increased mortality. Scholars van Oostrom et al. classified frailty into four types: physical frailty, psychological frailty, cognitive frailty, and social frailty. They also verified that sociodemographic factors, lifestyle, and multiple diseases affect the four types of frailty . In Taiwan, most frailty research focuses on the physiological aspects. Cognitive impairment and physical frailty are common health problems in the elderly, and the relationship between the two has been widely discussed. Many studies have confirmed that physical activity can not only reduce the occurrence of cognitive impairment but also is an important factor in reducing physiological frailty. The main reason is that physical activity can stimulate endothelial function and cell molecules in series, producing a protective mechanism to fight against cognitive decline and muscle loss. However, even though frailty and cognitive impairment are linked, the two conditions are often studied separately.

In recent years, domestic and foreign scholars have begun to realize the issues related to cognitive frailty (CF) and have begun to explore its prevalence, related influencing factors, influencing results, and intervention measures. According to the literature, the prevalence of cognitive frailty has increased significantly in recent years. The prevalence of cognitive impairment among community-dwelling older adults is 9% on average, with a prevalence of 13.3% in Taiwan. This increase in data is of great significance for the adjustment of health policies, nursing, and long-term care development. Literature shows that cognitive decline is a reversible state. If pay attention to this problem and start taking relevant intervention measures, we can avoid its rapid development.

The concept and assessment of cognitive decline in the elderly have been embryonic for the past five years. Conceptual definitions have been developed abroad. In recent years, many empirical studies have been conducted, most of which focus on longitudinal studies and dual-task intervention programs to verify the effects of cognitive function and physical activity on patients with cognitive impairment, but there is still a lack of randomized controlled trials. Although there are many studies on frailty in old adults in Taiwan, most of them are still Cognitive function, and physical frailty has been studied separately, and there are few studies on the topic of cognitive frailty. Therefore, this study introduced the cognitive-motor dual task of digital technology to understand the effectiveness of the dual task in cases of cognitive impairment.

Purpose:

1. Develop dual-task intervention solutions for digital technology.
2. To explore the effectiveness of dual-task intervention programs on cognitive function in older adults with cognitive impairment.
3. To explore the effectiveness of a dual-task intervention program on physical activity in cognitively impaired older adults.

Subjects:

1. Inclusion criteria: (1) aged 65 years or older; (2) subjective cognitive decline (measured by SMC with a score of at least 1 point) or mild cognitive impairment (measured by MoCA-T with a score of ≤25 points); (3) Possessing characteristics of physiological frailty (meeting at least one of the above items as measured by FFI).
2. Exclusion criteria: (1) diagnosed with Alzheimer's disease or other types of dementia; (2) suffering from musculoskeletal diseases and severe mental illness that make it impossible to perform cognitive and motor tasks.
3. Number of subjects: 50 in the experimental group and 50 in the control group
4. Recruitment method: (1) Recruitment location: residential institutions and senior citizen apartments in Taipei and New Taipei City (2) Recruitment through information sessions (with promotional posters)

Research design:

1. Study design or implementation This study used a randomized clinical trial to explore the effectiveness of a dual-task intervention program on cognitive function and physical activity in cognitively impaired older adults. This study was a single-blind, parallel randomized design, and the intervention began immediately after the initial evaluation and randomization. Eligible subjects were recruited by convenience sampling and subsequently randomly assigned to two groups: the experimental group received the dual-task regimen, and the control group received conventional care. The intervention activities of this study were cognitive and physical activity training using Nintendo Switch twice a week, 60 minutes each time (5 minutes of warm-up and cool-down exercises, 10 minutes of stretching exercises, and 40 minutes of exercise combined with cognitive training) for a total of 8 weeks. train. Both groups completed basic information (demographics and disease characteristics). They underwent cognitive function measurement at the pretest (T0), 4th week (T1), and 8th week (T2): the Taiwanese version of the Montreal Cognitive Assessment ( Taiwanese version of the Montreal Cognitive Assessment (MoCA-T), Trail Making Test (TMT), Taiwan Odd-Even Number Sequencing Test (TOENS); Physical activity function measurement: Timed Up and Test (Timed Up and Go, TUG), simple body measurement tool (Short Physical Performance Battery, SPPB) and handgrip strength test.
2. Project duration and expected progress

(1) This study was conducted after IRB and RCT were approved. (2) The case will be accepted after approval by both IRB and RCT. (3) Conduct data analysis and statistics after receiving the case 3. Statistical methods and results evaluation

1. Descriptive data analysis

   ①. Describe various demographic variables with frequency and percentage, including gender, marital status, education level, employment, living alone, economic status, chronic diseases, depression, dental and chewing function, medication use, physical activity (leisure sports), and Participation in social activities.

   ②. Describe continuous variables using mean, standard deviation, minimum, maximum, and range, including age, BMI, duration of illness, and medication use.
2. Inferential Data Analysis This study used an independent sample t-test and Chi-square test to detect the homogeneity of the two groups in terms of demographic variables, disease treatment variables, lifestyle habits, cognitive function, and physical activity. Since this study adopts a two-group (one before and two after) repeated measurement design, the generalized estimating equation (GEE) is used to handle repeated measurement data. Its advantages are that it allows the existence of missing values and assumes that Missing entirely at random (MACR) has the advantage of robust standard error and can handle continuous or binary variables. Therefore, GEE was used to analyze the intergroup effects of the two groups after dual-task intervention. And differences in the impact of between-group and time interactions.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Subjective cognitive decline (measured by SMC with a score of at least 1 point) or mild cognitive impairment (measured by MoCA-T with a score of ≤25 points)
* Possessing characteristics of physiological frailty (meeting at least one of the above items as measured by FFI)

Exclusion Criteria:

* Diagnosed with Alzheimer's disease or other types of dementia
* Suffering from musculoskeletal diseases and severe mental illness that make it impossible to perform cognitive and motor tasks

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Taiwanese version of the Montreal Cognitive Assessment (MoCA-T) | Baseline, pre-intervention (T0)
  This scale is used to assess the cognition funtion. The internal consistency Cronbach's coefficient of this tool is 0.83 and the test-retest reliability is 0.92.
Taiwanese version of the Montreal Cognitive Assessment (MoCA-T) | Four weeks after intervention(T1=4Weeks)
  This scale is used to assess the cognition funtion. The internal consistency Cronbach's coefficient of this tool is 0.83 and the test-retest reliability is 0.92.
Taiwanese version of the Montreal Cognitive Assessment (MoCA-T) | Eight weeks after intervention(T2=8Weeks)
  This scale is used to assess the cognition funtion. The internal consistency Cronbach's coefficient of this tool is 0.83 and the test-retest reliability is 0.92.
Taiwan Odd-Even Number Sequencing Test (TOENS) | Baseline, pre-intervention (T0)
  This scale is used to assess the cognition funtion. It's Half-reliability ranged from 0.69 to 0.95, and the test-retest reliability was 0.75.
Taiwan Odd-Even Number Sequencing Test (TOENS) | Four weeks after intervention(T1=4Weeks)
  This scale is used to assess the cognition funtion. It's Half-reliability ranged from 0.69 to 0.95, and the test-retest reliability was 0.75.
Taiwan Odd-Even Number Sequencing Test (TOENS) | Eight weeks after intervention(T2=8Weeks)
  This scale is used to assess the cognition funtion. It's Half-reliability ranged from 0.69 to 0.95, and the test-retest reliability was 0.75.
Trail Making Test (TMT) | Baseline, pre-intervention (T0)
  This scale is used to assess cognition function. The retest reliability of TMT-A is above 0.80 (0.60 ~0.90), and the retest reliability of TMT-B is 0.75
Trail Making Test (TMT) | Four weeks after intervention(T1=4Weeks)
  This scale is used to assess cognition function. The retest reliability of TMT-A is above 0.80 (0.60 ~0.90), and the retest reliability of TMT-B is 0.75
Trail Making Test (TMT) | Eight weeks after intervention(T2=8Weeks)
  This scale is used to assess cognition function. The retest reliability of TMT-A is above 0.80 (0.60 ~0.90), and the retest reliability of TMT-B is 0.75

SECONDARY OUTCOMES:
Timed Up and Go (TUG) | Baseline, pre-intervention (T0)
  This tool is used to assess physical activity function. The reliability of the tool is 0.96
Timed Up and Go (TUG) | Four weeks after intervention(T1=4Weeks)
  This tool is used to assess physical activity function. The reliability of the tool is 0.96
Timed Up and Go (TUG) | Eight weeks after intervention
  This tool is used to assess physical activity function. The reliability of the tool is 0.96
Short Physical Performance Battery (SPPB) | Baseline, pre-intervention (T0)
  This tool is used to assess physical activity function. The test-retest reliability of the SPPB was good: 0.87 (CI 95%: 0.77-0.96)
Short Physical Performance Battery (SPPB) | Four weeks after intervention(T1=4Weeks)
  This tool is used to assess physical activity function. The test-retest reliability of the SPPB was good: 0.87 (CI 95%: 0.77-0.96)
Short Physical Performance Battery (SPPB) | Eight weeks after intervention
  This tool is used to assess physical activity function. The test-retest reliability of the SPPB was good: 0.87 (CI 95%: 0.77-0.96)
Handgrip strength test | Baseline, pre-intervention (T0)
  This tool is used to assess physical activity function. This tool has been shown to be effective in research.
Handgrip strength test | Four weeks after intervention(T1=4Weeks)
  This tool is used to assess physical activity function. This tool has been shown to be effective in research.
Handgrip strength test | Eight weeks after intervention(T2=8Weeks)
  This tool is used to assess physical activity function. This tool has been shown to be effective in research.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruan Q, Yu Z, Chen M, Bao Z, Li J, He W. Cognitive frailty, a novel target for the prevention of elderly dependency. Ageing Res Rev. 2015 Mar;20:1-10. doi: 10.1016/j.arr.2014.12.004. Epub 2014 Dec 30. PMID 25555677
- [Background] Qiu Y, Li G, Wang X, Zheng L, Wang C, Wang C, Chen L. Prevalence of cognitive frailty among community-dwelling older adults: A systematic review and meta-analysis. Int J Nurs Stud. 2022 Jan;125:104112. doi: 10.1016/j.ijnurstu.2021.104112. Epub 2021 Oct 18. PMID 34758429
- [Background] van Oostrom SH, van der A DL, Rietman ML, Picavet HSJ, Lette M, Verschuren WMM, de Bruin SR, Spijkerman AMW. A four-domain approach of frailty explored in the Doetinchem Cohort Study. BMC Geriatr. 2017 Aug 30;17(1):196. doi: 10.1186/s12877-017-0595-0. PMID 28854882
- [Background] Mantovani E, Zucchella C, Schena F, Romanelli MG, Venturelli M, Tamburin S. Towards a Redefinition of Cognitive Frailty. J Alzheimers Dis. 2020;76(3):831-843. doi: 10.3233/JAD-200137. PMID 32568197
- [Background] Lauretani F, Longobucco Y, Ferrari Pellegrini F, De Iorio AM, Fazio C, Federici R, Gallini E, La Porta U, Ravazzoni G, Roberti MF, Salvi M, Zucchini I, Pela G, Maggio M. Comprehensive Model for Physical and Cognitive Frailty: Current Organization and Unmet Needs. Front Psychol. 2020 Nov 26;11:569629. doi: 10.3389/fpsyg.2020.569629. eCollection 2020. PMID 33324282
- [Background] Kwan RYC, Liu JYW, Fong KNK, Qin J, Leung PK, Sin OSK, Hon PY, Suen LW, Tse MK, Lai CK. Feasibility and Effects of Virtual Reality Motor-Cognitive Training in Community-Dwelling Older People With Cognitive Frailty: Pilot Randomized Controlled Trial. JMIR Serious Games. 2021 Aug 6;9(3):e28400. doi: 10.2196/28400. PMID 34383662
- [Background] Kwan RY, Lee D, Lee PH, Tse M, Cheung DS, Thiamwong L, Choi KS. Effects of an mHealth Brisk Walking Intervention on Increasing Physical Activity in Older People With Cognitive Frailty: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Jul 31;8(7):e16596. doi: 10.2196/16596. PMID 32735218
- [Background] Kelaiditi E, Cesari M, Canevelli M, van Kan GA, Ousset PJ, Gillette-Guyonnet S, Ritz P, Duveau F, Soto ME, Provencher V, Nourhashemi F, Salva A, Robert P, Andrieu S, Rolland Y, Touchon J, Fitten JL, Vellas B; IANA/IAGG. Cognitive frailty: rational and definition from an (I.A.N.A./I.A.G.G.) international consensus group. J Nutr Health Aging. 2013 Sep;17(9):726-34. doi: 10.1007/s12603-013-0367-2. PMID 24154642
- [Background] Junius-Walker U, Onder G, Soleymani D, Wiese B, Albaina O, Bernabei R, Marzetti E; ADVANTAGE JA WP4 group. The essence of frailty: A systematic review and qualitative synthesis on frailty concepts and definitions. Eur J Intern Med. 2018 Oct;56:3-10. doi: 10.1016/j.ejim.2018.04.023. Epub 2018 May 31. PMID 29861330
- [Background] Jiayuan Z, Xiang-Zi J, Li-Na M, Jin-Wei Y, Xue Y. Effects of Mindfulness-Based Tai Chi Chuan on Physical Performance and Cognitive Function among Cognitive Frailty Older Adults: A Six-Month Follow-Up of a Randomized Controlled Trial. J Prev Alzheimers Dis. 2022;9(1):104-112. doi: 10.14283/jpad.2021.40. PMID 35098980